CLINICAL TRIAL: NCT02063217
Title: Modulation of CSF Amyloid-beta Concentrations Via Behavioral Sleep Deprivation and Pharmacological Sleep Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201304030; P50AG005681-30 (NIH)
Record Dates: First submitted 2014-01-29; First posted 2014-02-14 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-04-26 (Actual); Status verified 2018-03

CONDITIONS: Amyloid-beta
MeSH Terms: conditions — Plaque, Amyloid | interventions — Sodium Oxybate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sleep Induction (Experimental): 7.5 grams of sodium oxybate
  Interventions: Drug: Sodium Oxybate
- Sleep Deprivation (Experimental): Sleep deprivation for up to 36 hours with no naps or other sleep periods
  Interventions: Behavioral: Sleep deprivation
- Control (No Intervention): Participant will sleep as normal under the same controlled conditions in a clinical research unit

INTERVENTIONS:
Drug: Sodium Oxybate — Sodium oxybate h.s.
  Other Names: Xyrem
  Arms: Sleep Induction
Behavioral: Sleep deprivation — 36hr sleep deprivation
  Arms: Sleep Deprivation

SUMMARY:
The purpose of this study is to change the concentration of amyloid-beta in human cerebrospinal fluid (CSF) through modulation of the sleep-wake cycle.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate whether or not increasing or decreasing duration of sleep over one night will change the concentration of amyloid-beta in cerebral spinal fluid (CSF).

ELIGIBILITY:
Inclusion Criteria:

* cognitively normal or CDR 0
* negative for amyloid deposition by PET Pittsburgh Compound-B (PIB) imaging or CSF amyloid-beta-42 concentration
* Age 18-60
* Average reported sleep time 6-10hrs

Exclusion Criteria:

* diagnosis of a sleep disorder such as sleep apnea, narcolepsy, or restless leg syndrome
* positive ambulatory sleep study for obstructive sleep apnea (AHI > 5 respiratory events per hour) that will be performed as part of initial screening prior to enrollment
* Clinical Dementia Rating (CDR) > 0
* tremor or other neurologic injury in the non-dominant upper extremity (such as stroke or tremor) that would prevent the use of actigraphy
* current sleep walking or other sleep parasomnia
* diagnosis and treatment of stroke, myocardial infarction or heart attack,
* coronary artery disease, atrial fibrillation, or congestive heart failure
* diagnosis and treatment of asthma or Chronic Obstructive Pulmonary Disease (COPD)
* diagnosis and treatment of bipolar disorder, major depression, or Schizophrenia
* current urinary or fecal incontinence
* currently on a low salt diet
* diagnosis and treatment of a neurologic disorder such as Parkinson's disease, epilepsy, multiple sclerosis
* currently taking any blood thinner medications such as warfarin, Plavix, or Aspirin
* kidney disease resulting in renal impairment
* liver disease resulting in hepatic dysfunction
* Pregnancy
* currently taking sedating medications such as benzodiazepines
* alcohol use at bedtime
* tobacco use
* BMI >40
* contraindication to lumbar puncture
* diabetes
* sleep schedule outside the range of bedtime: 8pm-12am and waketime 4am-8am
* self reported difficulty sleeping in an unfamiliar environment
* use of sedative-hypnotic medications
* inability to get in and out of bed
* history or presence of any clinically significant medical condition, behavioral or psychiatric disorder, or surgical history based on medical record or patient report
* history of drug abuse within the past 6 months
* positive score on 2 or more categories on the Berlin questionnaire
* participation in another investigational medicinal product or investigational device within the last 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-12; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lucey, MD, Principal Investigator — Washington University Medical School
Locations (1):
- Washington University Medical School, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sleep Induction: 6.5-7.5 grams of sodium oxybate
  Sodium Oxybate: Sodium oxybate h.s.
Period: Overall Study
Arm/Group | Sleep Induction | Sleep Deprivation | Control
Started | 12 | 12 | 12
Completed (All participants invited to repeat the study; enrollment totals include repeat participants.) | 11 | 12 | 12
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Induction | Sleep Deprivation | Control | Total
Number analyzed (Participants) | 11 | 12 | 12 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 12 | 35
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 45.5 [20.8 to 58.3] | 42.0 [18.8 to 58.6] | 42.7 [25 to 57.2] | 43.3 [18.8 to 58.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 8 | 19
  Male | 6 | 6 | 4 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 12 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percent Increase From Mean Baseline (07:00 to 19:00) of Cerebrospinal Fluid (CSF) Amyloid Beta During Sleep Induction and Sleep Deprivation Between 01:00 and 11:00 From Baseline
Description: Overnight (01:00 to 11:00) differences in CSF amyloid beta from baseline (07:00 to 19:00) between 1) sleep-deprived and control participants and 2) sleep-induced and control participants.
Time Frame: Baseline = 07:00 to 19:00; Intervention period = 01:00 to 11:00
Population: Participants in good general health who had CSF collected every 2 hours for 36 hours while undergoing with sleep deprivation, sleep induction with drug, or control conditions.
Measure: Mean (Standard Error); unit: percent increase from mean baseline
Arm/Group | Sleep Induction | Sleep Deprivation | Control
Number analyzed (Participants) | 11 | 12 | 12
percent increase from mean baseline | 113 (5.7) | 123 (6.6) | 106 (5.6)
Statistical Analysis 1: Comparison: Sleep Deprivation vs Control; Mixed linear modeling of change in overnight amyloid beta concentrations from waking baseline between 01:00 and 11:00. Data provided for amyloid beta-40; Test type: Superiority — Mixed linear models; p = 0.07, Mixed Models Analysis — Bonferroni correction was used for multiple comparisons; Mean Difference (Net) = 17 — Mean (standard error), units = %. 17(7.2) increase in overnight amyloid-beta 40 concentrations over waking baseline between the sleep deprivation group and controls
Statistical Analysis 2: Comparison: Sleep Induction vs Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — Mixed linear models; p = 1.0, Mixed Models Analysis — Bonferroni correction was used for multiple comparisons; Mean Difference (Net) = 7 — Mean= 7%, standard error = 7.6%. 7% increase in overnight amyloid beta 40 concentrations over the waking baseline between the sleep induction group and control group

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the start of the participant confinement visits to the Clinical Research Unit when the lumbar catheter was placed and cerebrospinal fluid collected. Adverse event recording continued through a 48 hour telephone follow-up period. Total reporting period was 6 days.
Arm/Group | Sleep Induction | Sleep Deprivation | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 11/12 | 9/12 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sleep Induction (N=12) | Sleep Deprivation (N=12) | Control (N=12)
Headache (Nervous system disorders) | 10 (10) | 8 (8) | 8 (8)
Headache requiring blood patch (Nervous system disorders) | 4 (4) | 4 (4) | 0 (0) — Headache requiring blood patch after removal of the lumbar catheter.
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 1 (1)
Presyncope/syncope with lumbar catheter placement (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Leg tingling (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Back/neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) — Back/neck pain requiring acetaminophen
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sweating (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No